CLINICAL TRIAL: NCT03145285
Title: Activity of Abiraterone Acetate in the Management of Cushing's Syndrome in Patients With Adrenocortical Carcinoma
Acronym: ABACUS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Niguarda Hospital (Other); San Camillo Hospital, Rome (Other); San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Salvatore Grisanti, MD, PhD, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASSTBS-ONCO-ABACUS-16; 2016-000945-29 (EudraCT Number)
Record Dates: First submitted 2017-04-26; First posted 2017-05-09 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Cushing Syndrome; Adrenocortical Carcinoma
Keywords: Abiraterone Acetate; Cushing Syndrome; Adrenocortical Carcinoma
MeSH Terms: conditions — Cushing Syndrome; Adrenocortical Carcinoma | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Patients locally advanced/metastatic ACC patients with uncontrolled Cushing's syndrome despite Mitotane +/- chemotherapy.
  Treatment with single agent Abiraterone Acetate (AA) until progression
  Interventions: Drug: Abiraterone Acetate
- Cohort 2 (Experimental): Mitotane-naïve patients with newly diagnosis of ACC associated with Cushing's syndrome not amenable to surgical resection.
  Treatment with single agent Abiraterone Acetate (AA) for 4 weeks followed by AA + Mitotane +/- first-line chemotherapy. AA in association with Mitotane will be administered for 3 months. If the primary endpoint is obtained before 1 month, then Mitotane +/- chemotherapy can be started upon the clinician's decision.
  Interventions: Drug: Abiraterone Acetate

INTERVENTIONS:
Drug: Abiraterone Acetate — Cohort 1:
  Patients locally advanced/metastatic ACC patients with uncontrolled Cushing's syndrome despite Mitotane +/- chemotherapy will be treated with single agent AA.Mitotane and chemotherapy will be interrupted and AA will be continued till progression and/or until progression of Cushing's syndrome.
  Cohort 2:
  Mitotane-naïve patients with newly diagnosis of ACC associated with Cushing's syndrome not amenable to surgical resection will be treated with AA for 4 weeks followed by AA + Mitotane +/- first-line chemotherapy. AA in association with Mitotane will be administered for 3 months. If the primary endpoint is obtained before 1 month (i.e. 2 or 3 weeks from Abiraterone start), then Mitotane +/- chemotherapy can be started upon the clinician's decision.
  Other Names: Zytiga

SUMMARY:
Adrenocortical Carcinoma (ACC) is an extremely rare disease. Approximately 50% of ACC in adults are functioning leading to hormonal and metabolic syndromes. Cortisol hypersecretion (Cushing's syndrome) is the most common endocrine derangement at presentation. Moreover, hypercortisolism is one of the factors that negatively influence the outcome of patients with metastatic ACC.

Abiraterone acetate (AA) is a prodrug of abiraterone, an irreversible inhibitor of 17α hydroxylase/C17, 20-lyase (cytochrome P450c17 [CYP17]).The inhibition of CYP17A1 blocks androgen and cortisol synthesis. AA has a pharmacodynamic potential to reduce cortisol excess and it has never been tested before in Cushing's syndrome.

Thus, we decided to evaluate the activity of Abiraterone Acetate in the management of Cushing's syndrome in patients with adrenocortical carcinoma. The study is a phase II, non-randomized, open-label study with two different experimental sub-cohorts:

Cohort 1: Patients locally advanced/metastatic ACC patients with uncontrolled Cushing's syndrome despite Mitotane +/- chemotherapy will be treated with single agent AA. In this cohort, Mitotane and chemotherapy will be interrupted and AA will be continued till progression and/or as long as the Cushing's syndrome is adequately controlled (ie until progression of Cushing's syndrome).

Cohort 2: Mitotane-naïve patients with newly diagnosis of ACC associated with Cushing's syndrome not amenable to surgical resection with radical intent will be treated with single agent AA for 4 weeks followed by AA + Mitotane +/- first-line chemotherapy. In this cohort, AA in association with Mitotane will be administered for 3 months. If the primary endpoint is obtained before 1 month (i.e. 2 or 3 weeks from Abiraterone start), then Mitotane +/- chemotherapy can be started upon the clinician's decision.

DETAILED DESCRIPTION:
Background:

ACC is an extremely rare disease. About 30% of patients are diagnosed with locally/advanced metastatic disease and about 50-80% of patients who undergo radical resection are destined to relapse often with distant metastases. Approximately 50% of ACC in adults are functioning leading to hormonal and metabolic syndromes. Cortisol hypersecretion (Cushing's syndrome) is the most common endocrine derangement at presentation. Control of the syndrome is mainly obtained by mitotane therapy, however this drug requires several weeks to months for attaining a therapeutic range of serum concentrations. Hypercortisolism is one of the factors that negatively influence the outcome of patients with metastatic ACC.

Abiraterone acetate (AA) is a prodrug of abiraterone, an irreversible inhibitor of 17α hydroxylase/C17, 20-lyase (cytochrome P450c17 [CYP17]), that are key enzymes required for testosterone synthesis. These enzymes are found in the testes, adrenals and prostate tumors. The inhibition of CYP17A1 blocks androgen and cortisol synthesis. Abiraterone has demonstrated to be able to suppress dehydroepiandrosterone (DHEA), androstenedione and testosterone production in both adrenal and testes and to reduce adrenal cortisol production. For these reasons Abiraterone is registered for clinical use in castrate-resistant prostate cancer (CRPC). The maximum inhibition of CYP17A1 is achieved within 28 days of continuous dosing.

Rationale:

* A rapid control of the Cushing's syndrome is important in patients with ACC.
* AA has a pharmacodynamic potential to reduce cortisol excess and it has never been tested before in Cushing's syndrome.

Statistical considerations:

The sample size in Cohort 1 according to an Intent To Treat (ITT) procedure is calculated under the following considerations:

H0: current therapies can normalize UFC in 40% of patients in 1 month of therapy; H1: Abiraterone can normalize UFC in at least 70% of patients in 1 month of therapy.

Therefore, the sample size calculation is based on the comparison between the response observed with traditional therapies (R0 = 0.4) and the response expected with the experimental drug (R1 = 0.7). With a two-sided Chi-square test, twenty consecutive patients should be enrolled to detect a 30% absolute difference with an alpha error 5% and a power of 80%.

Considering the exploratory purpose of Cohort 2 substudy, no sample size has been determined and a total of 10 patients will be enrolled.

Abiraterone administration and dose modifications:

Abiraterone Acetate will be administered per os at the standard dose of four 250 mg capsules (1000 mg total dose) daily on an empty stomach in 28-day cycles.

In case of an adverse event (AE) where according to investigator judgement a dose-reduction is required, 1 dose reduction is allowed to 500 mg Abiraterone (4→2 tablets). Any return to protocol dose level (4 tablets) after dose reduction must follow documentation of adverse event resolution.

Safety and management of AEs:

The evaluation period for safety will start from signing of the informed consent form to at least 30 days after the last dose of study drug or recovery from all acute toxicities associated with study drug administration. Adverse events including laboratory AEs will be graded and summarized according to the NCI-CTCAE, Version 4.0. The study will include evaluations of safety according to the time points provided in the Time and Events Schedule.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diagnosis of ACC
* CT or MRI evidence of metastatic or locally advanced ACC (ENSAT stage III-IV) unsuitable for radical surgery
* Age ≥ 18 years
* Confirmed diagnosis of Cushing's syndrome validated by:
* two 24 h urinary collections for UFC at least 1.5 times the upper the normal levels, within 2 weeks prior to enrollment;
* serum ACTH levels lower than the normal range;
* ECOG performance status ≤ 2
* Effective contraception
* Patients must provide verbal and written informed consent to be enrolled in the study

Exclusion Criteria:

* Life expectancy less than 3 months
* Liver disease, such as cirrhosis, chronic or persistent active hepatitis or AST/ALT > 2 x ULN, bilirubin >2 x ULN
* Heart failure (NYHA class III or IV), unstable angina, severe arrhythmia or clinically significant impairment of heart function
* Major surgical procedure within one month prior entering the study
* Renal impairment (creatinine clearance < 40 ml/min).
* WBC <3 x 109 /L; Hb <13 g/dL for men and <12 g/dL for women; platelets <100 x 109 /L
* Any other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Pregnant or breast-feeding women
* History of alcohol or drug abuse
* History of recent or active prior malignancy, except for cured non-melanoma skin cancer, cured in situ cervical carcinoma, or other treated malignancies with no evidence of disease for at least three years)
* Acute or chronic uncontrolled infections
* Patient non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2020-04-18 (Estimated); Study Completion 2021-04-18 (Estimated)

PRIMARY OUTCOMES:
To assess the activity of AA in attaining normalization of 24-h urinary free cortisol (UFC) excretion relative to baseline within 1 month from treatment start | 1 month
  laboratory tests

SECONDARY OUTCOMES:
to assess the activity of AA in attaining 50% reduction of 24-h UFC excretion within 1 month of treatment | 1 month
  laboratory tests
time to reduction of UFC (compared to screening values) | Weekly, from date of treatment start, for the first month; thereafter every 2 months up to 48 months.
  laboratory tests (24-h UFC excretion)
effect of AA on levels of serum cortisol, UFC, salivary cortisol, ACTH, aldosterone, PRA, DHEA-S, total testosterone, and steroid precursors | Monthly, from date of treatment start, for the first 3 months; thereafter every 2 months up to 48 months
  laboratory tests
improvement of the clinical signs associated to hypercortisolism | every visit up to 48 months
  multiparameter scoring based on clinical signs/and symptoms and biochemical alterations associated to hypercortisolism
improvement of quality of life | every visit up to 48 months
  evaluation of validated questionnaire (FACT-G)
safety and tolerability of oral assumption of AA | Weekly, from date of treatment start, for the first month; once a month for the first 3 months; thereafter every 2 months up to 48 months
  evaluation of side effects appearance with study drug using the National Cancer Institute Common Toxicity Criteria (NCI-CTCAE)
treatment response (according to RECIST criteria) | every 3 months or earlier upon clinician's decision, up to 48 months
  CT total body or MRI scan or FDG PET
progression-free survival | every visit up to 48 months
  defined as the time elapsing from patient registration to first evidence of disease progression
time to syndrome relapse | every visit up to 48 months
  defined as the time elapsing from the best syndrome control within the first month to relapse of syndrome defined as: 1) Cushing symptoms recurrence; 2) increase more than 50% of nadir cortisol levels
overall survival | every visit up to 48 months
  defined as months from the first day of drug administration to the end of follow up or patient's death

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Grisanti, MD, PhD, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- U.O Oncologia Medica, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berruti A, Baudin E, Gelderblom H, Haak HR, Porpiglia F, Fassnacht M, Pentheroudakis G; ESMO Guidelines Working Group. Adrenal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2012 Oct;23 Suppl 7:vii131-8. doi: 10.1093/annonc/mds231. No abstract available. PMID 22997446
- [Result] Abiven G, Coste J, Groussin L, Anract P, Tissier F, Legmann P, Dousset B, Bertagna X, Bertherat J. Clinical and biological features in the prognosis of adrenocortical cancer: poor outcome of cortisol-secreting tumors in a series of 202 consecutive patients. J Clin Endocrinol Metab. 2006 Jul;91(7):2650-5. doi: 10.1210/jc.2005-2730. Epub 2006 May 2. PMID 16670169
- [Result] Berruti A, Terzolo M, Sperone P, Pia A, Della Casa S, Gross DJ, Carnaghi C, Casali P, Porpiglia F, Mantero F, Reimondo G, Angeli A, Dogliotti L. Etoposide, doxorubicin and cisplatin plus mitotane in the treatment of advanced adrenocortical carcinoma: a large prospective phase II trial. Endocr Relat Cancer. 2005 Sep;12(3):657-66. doi: 10.1677/erc.1.01025. PMID 16172198
- [Result] Berruti A, Fassnacht M, Haak H, Else T, Baudin E, Sperone P, Kroiss M, Kerkhofs T, Williams AR, Ardito A, Leboulleux S, Volante M, Deutschbein T, Feelders R, Ronchi C, Grisanti S, Gelderblom H, Porpiglia F, Papotti M, Hammer GD, Allolio B, Terzolo M. Prognostic role of overt hypercortisolism in completely operated patients with adrenocortical cancer. Eur Urol. 2014 Apr;65(4):832-8. doi: 10.1016/j.eururo.2013.11.006. Epub 2013 Nov 14. PMID 24268504
- [Result] Daniel E, Aylwin S, Mustafa O, Ball S, Munir A, Boelaert K, Chortis V, Cuthbertson DJ, Daousi C, Rajeev SP, Davis J, Cheer K, Drake W, Gunganah K, Grossman A, Gurnell M, Powlson AS, Karavitaki N, Huguet I, Kearney T, Mohit K, Meeran K, Hill N, Rees A, Lansdown AJ, Trainer PJ, Minder AE, Newell-Price J. Effectiveness of Metyrapone in Treating Cushing's Syndrome: A Retrospective Multicenter Study in 195 Patients. J Clin Endocrinol Metab. 2015 Nov;100(11):4146-54. doi: 10.1210/jc.2015-2616. Epub 2015 Sep 9. PMID 26353009
- [Result] Dharia S, Slane A, Jian M, Conner M, Conley AJ, Parker CR Jr. Colocalization of P450c17 and cytochrome b5 in androgen-synthesizing tissues of the human. Biol Reprod. 2004 Jul;71(1):83-8. doi: 10.1095/biolreprod.103.026732. Epub 2004 Feb 25. PMID 14985252
- [Result] de Bono JS, Logothetis CJ, Molina A, Fizazi K, North S, Chu L, Chi KN, Jones RJ, Goodman OB Jr, Saad F, Staffurth JN, Mainwaring P, Harland S, Flaig TW, Hutson TE, Cheng T, Patterson H, Hainsworth JD, Ryan CJ, Sternberg CN, Ellard SL, Flechon A, Saleh M, Scholz M, Efstathiou E, Zivi A, Bianchini D, Loriot Y, Chieffo N, Kheoh T, Haqq CM, Scher HI; COU-AA-301 Investigators. Abiraterone and increased survival in metastatic prostate cancer. N Engl J Med. 2011 May 26;364(21):1995-2005. doi: 10.1056/NEJMoa1014618. PMID 21612468
- [Result] Trump DL. Commentary on "Abiraterone in metastatic prostate cancer without previous chemotherapy." Ryan CJ, Smith MR, de Bono JS, Molina A, Logothetis CJ, de Souza P, Fizazi K, Mainwaring P, Piulats JM, Ng S, Carles J, Mulders PF, Basch E, Small EJ, Saad F, Schrijvers D, Van Poppel H, Mukherjee SD, Suttmann H, Gerritsen WR, Flaig TW, George DJ, Yu EY, Efstathiou E, Pantuck A, Winquist E, Higano CS, Taplin ME, Park Y, Kheoh T, Griffin T, Scher HI, Rathkopf DE; COU-AA-302 Investigators, Genitourinary Medical Oncology Program, Helen Diller Family Comprehensive Cancer Center, University of California, San Francisco, CA. N Engl J Med 2013;368(2):138-48 [Epub 2012 Dec 10]; N Engl J Med 2013;368(6):584. Urol Oncol. 2013 Nov;31(8):1846. doi: 10.1016/j.urolonc.2013.08.012. PMID 24210085
- [Result] Ang JE, Olmos D, de Bono JS. CYP17 blockade by abiraterone: further evidence for frequent continued hormone-dependence in castration-resistant prostate cancer. Br J Cancer. 2009 Mar 10;100(5):671-5. doi: 10.1038/sj.bjc.6604904. Epub 2009 Feb 17. PMID 19223900
- [Result] Yap TA, Carden CP, Attard G, de Bono JS. Targeting CYP17: established and novel approaches in prostate cancer. Curr Opin Pharmacol. 2008 Aug;8(4):449-57. doi: 10.1016/j.coph.2008.06.004. Epub 2008 Jul 28. PMID 18619560
- [Result] Krone N, Arlt W. Genetics of congenital adrenal hyperplasia. Best Pract Res Clin Endocrinol Metab. 2009 Apr;23(2):181-92. doi: 10.1016/j.beem.2008.10.014. PMID 19500762
- [Result] Ferraldeschi R, Sharifi N, Auchus RJ, Attard G. Molecular pathways: Inhibiting steroid biosynthesis in prostate cancer. Clin Cancer Res. 2013 Jul 1;19(13):3353-9. doi: 10.1158/1078-0432.CCR-12-0931. Epub 2013 Mar 7. PMID 23470964
- [Result] Baudin E, Pellegriti G, Bonnay M, Penfornis A, Laplanche A, Vassal G, Schlumberger M. Impact of monitoring plasma 1,1-dichlorodiphenildichloroethane (o,p'DDD) levels on the treatment of patients with adrenocortical carcinoma. Cancer. 2001 Sep 15;92(6):1385-92. doi: 10.1002/1097-0142(20010915)92:63.0.co;2-2. PMID 11745214
- [Result] van Erp NP, Guchelaar HJ, Ploeger BA, Romijn JA, Hartigh Jd, Gelderblom H. Mitotane has a strong and a durable inducing effect on CYP3A4 activity. Eur J Endocrinol. 2011 Apr;164(4):621-6. doi: 10.1530/EJE-10-0956. Epub 2011 Jan 10. PMID 21220434
- [Result] Chung E, Nafziger AN, Kazierad DJ, Bertino JS Jr. Comparison of midazolam and simvastatin as cytochrome P450 3A probes. Clin Pharmacol Ther. 2006 Apr;79(4):350-61. doi: 10.1016/j.clpt.2005.11.016. Epub 2006 Feb 28. PMID 16580903